CLINICAL TRIAL: NCT01195454
Title: Euglycemic Clamp Dose-response Study Comparing a New Insulin Glargine Formulation With Lantus®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PKD11627; 2010-020914-27 (EudraCT Number)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin glargine / New insulin glargine formulation (Experimental): * Period 1: Insulin glargine
  * Period 2: New insulin glargine formulation
  * Period 3: New insulin glargine formulation
  * Period 4: New insulin glargine formulation
  Duration of treatment: 1 day at each period
  Interventions: Drug: Insulin glargine (HOE901)

INTERVENTIONS:
Drug: Insulin glargine (HOE901) — Pharmaceutical form: Lantus solution for injection
  Route of administration: subcutaneous
Drug: Insulin glargine (HOE901) — Pharmaceutical form: New insulin glargine formulation solution for injection
  Route of administration: subcutaneous

SUMMARY:
Primary Objective:

- To assess the total metabolic effect ratios of a new insulin glargine formulation versus Lantus®

Secondary Objectives:

* To assess the exposure ratios of a new insulin glargine formulation versus Lantus®
* To compare the duration of action of a new insulin glargine formulation versus Lantus®
* To explore the dose response and dose exposure relationship of a new insulin glargine formulation
* To assess the safety and tolerability of a new insulin glargine formulation

DETAILED DESCRIPTION:
The study period for one patient is one month in average and it can last up to 11 weeks broken down as follows:

* Screening: 3 to 28 days
* Treatment period: 1 to 4 days: 2 days (1 overnight stay)
* Washout period: 5 to 18 days (preferentially 7 days between consecutive dosings)
* End of study: 1 day after the last dosing

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects with diabetes mellitus type 1 for more than one year,
* Total insulin dose of <1.2 U/kg/day,
* Glycohemoglobin (HbA1c) ≤ 9.0%,
* Fasting negative serum C-peptide (< 0.3 nmol/L),
* Stable insulin regimen for at least 2 months prior to study,
* Normal findings in medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and musculo-skeletal system), vital signs, electrocardiogram (ECG) and safety lab,
* Women of childbearing potential with negative pregnancy test and use of a highly effective contraceptive method or women with confirmed postmenopausal status.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic (apart from diabetes mellitus type 1), hematological, neurological, psychiatric, systemic (affecting the body as a whole), ocular, gynecologic (if female), or infectious disease; any acute infectious disease or signs of acute illness,
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months,
* Frequent severe headaches and / or migraine, recurrent nausea and / or vomiting (more than twice a month),
* Symptomatic hypotension (whatever the decrease in blood pressure), or asymptomatic postural hypotension defined by a decrease in SBP equal to or greater than 20 mmHg within three minutes when changing from the supine to the standing position,
* Presence or history of a drug allergy or clinically significant allergic disease,
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol,
* Pregnant or breast feeding women,
* Any medication (including St John's Wort) within 14 days before inclusion, or within 5 times the elimination half-life or pharmacodynamic half-life of that drug, whichever the longest and regular use of any medication other than insulins in the last month before study start with the exception of thyroid hormones, lipid-lowering and antihypertensive drugs, and, if female, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days,
* Positive reaction to any of the following tests: hepatitis B surface (HBs Ag) antigen, antihepatitis B core antibodies (anti-HBc Ab) if compound having possible immune activities, anti-hepatitis C virus (anti-HCV2) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab),
* Known hypersensitivity to insulin glargine and excipients,
* Any history or presence of deep leg vein thrombosis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The area under the body weight standardized glucose infusion rate curve (GIR) within 36 hours (GIR-AUC0-36) | 36 hours (D1 to D2) in all four treatment periods

SECONDARY OUTCOMES:
The area under the insulin glargine concentration curve within 36 hours (INS-AUC0-36) - | 36 hours (D1 to D2) in all four treatment periods
Time to 50% of the GIR-AUC0-36 (T50%-GIR AUC0-36) | 36 hours (D1 to D2) in all four treatment periods
Time to 50% of INS-AUC0-36 (T50% INS-AUC0-36) | 36 hours (D1 to D2) in all four treatment periods
Duration of blood glucose control (time to elevation of smoothed blood glucose profile above clamp level and to elevation above different pre-specified blood glucose levels) | 36 hours (D1 to D2) in all four treatment periods
Maximum smoothed body weight standardized glucose infusion rate GIRmax, and time to GIRmax (GIR-Tmax) | 36 hours (D1 to D2) in all four treatment periods
Maximum insulin concentration INS-Cmax, and time to Cmax (INS-Tmax) | 36 hours (D1 to D2) in all four treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Berlin, Germany